CLINICAL TRIAL: NCT06026306
Title: A Pilot Randomized Controlled Trial of a Scalable Psychological Intervention for Enhancing Mental Health Outcomes Among Earthquake Survivors in Türkiye
Brief Title: A Scalable Psychological Intervention for Earthquake Survivors in Türkiye
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023.271.IRB3.125
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-08

CONDITIONS: Psychological Distress; Impaired Social Functioning; Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants will not be blinded to their study arm because of the nature of the intervention, but outcome assessors will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Problem Management Plus (PM+) (Experimental): The experimental group will receive a 5-session individual PM+.
  Interventions: Behavioral: Problem Management Plus (PM+)
- Enhanced Care as Usual (No Intervention): The control (enhanced care as usual) group will receive the information about freely available psychological support options. E-CAU ranges from standard community care which may include any existing mental health support services available to earthquake survivors in container cities. The participants will be given flyers which include information about the services provided by the government and by non-governmental organizations. After completion of the post and follow-up assessment of experimental group, those in the E-CAU condition will be offered with PM+.

INTERVENTIONS:
Behavioral: Problem Management Plus (PM+) — PM+ consists of five weekly in-person sessions of 90 minutes. The intervention integrates four evidence-based behavioural strategies: arousal reduction using a slow breathing exercise (session 1), problem-solving (session 2), behavioural activation by re-engaging with pleasant and task-oriented activities (session 3) and accessing social support (session 4). Homework practice is scheduled following each session and discussed in the next session. Psychoeducation is delivered in session 1 and relapse prevention is discussed in session
  Arms: Problem Management Plus (PM+)

SUMMARY:
This will be the first pilot randomized controlled trial (RCT) study that investigate the potential effectiveness of individual PM+ among earthquake survivors residing in container cities in Türkiye. The primary objective of this pilot study will be to test feasibility, acceptability, and potential effectiveness of individual PM+ for Turkish earthquake survivors, using RCT design which is considered the gold standard in research for evaluating effectiveness of interventions. Secondly, this study aims to test trial procedures in preparation for a future larger randomized controlled trial.

DETAILED DESCRIPTION:
On the 6th February, 2023, Türkiye experienced two consecutive earthquakes with magnitudes of 7.7 and 7.6. As a consequence of such a disaster, the increasing prevalence of mental health issues has resulted in increased need and demand for mental health and psychosocial support (MHPSS) services in the country. In order to reach a higher number of people on time, implementation of brief, scalable interventions addressing common mental health problems has garnered significant importance. One such intervention is Problem Management Plus that is developed by World Health Organization for communities that experienced adversities. PM+ is a 5-session psychological intervention that aims to improve common mental health problems by teaching participants evidence-based behavioral strategies (i.e., stress management, problem solving, behavioral activation and strengthening social support). Both the individual and group versions of PM+ were tested for feasibility, acceptability, and effectiveness in various countries among different populations, including the earthquake-affected communities in Nepal.

This study will be the first to test the potential effectiveness of individual PM+ among earthquake survivors in Türkiye. The study will be designed as a pilot randomized controlled trial and the potential effectiveness of individual PM+ will be tested compared to Enhanced-Care as Usual (E-CAU) control group. The study is planned to be conducted at container cities in different earthquake regions (e.g.,Hatay, Adıyaman or Malatya). After the baseline assessment, eligible 60 participants will be randomized to two arms: in either the PM+ (n=30) or only control group (E-CAU; n=30). If they will be randomized into the PM+ condition, the facilitator will plan five consecutive sessions with the participants. The first session will take place no longer than one week after the pre-intervention assessment. The post-intervention assessment through the same measures used in the pretest will take place within 1 week after completion of the fifth session. Follow-up assessment will be conducted one month after the last-session. All study participants including drop-outs will be invited to all outcome assessments. After completion of the follow-up assessment, those in the E-CAU condition will be offered with PM+. The primary outcome measure will be depression and anxiety, posttraumatic stress, psychological distress, psychosocial functioning and self-identified problems will be included as secondary outcome measures.

In order to assess feasibility and acceptability of these interventions, and the possibility of scaling up as well, we will assess the recruitment and consent rates, the percentages of attendance of sessions, the protocol adherence, drop-out rates and qualitative assessments from the process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or above
* Being experienced the Kahramanmaraş earthquake
* Elevated level of psychological distress indicated by having a score of 15 or above on Kessler Psychological Distress Scale (K10)
* Impaired daily functioning indicated by having a score of 16 or above on WHO Disability Assessment Schedule (WHODAS)

Exclusion Criteria:

* imminent suicide risk (assessed with the PM+ manual suicidal thoughts interview),
* indications of severe mental disorders (e.g., psychotic disorders) or cognitive impairment (e.g., severe intellectual disability; assessed by the PM+ manual observation checklist),
* ongoing treatment in specialized mental health care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change of the Patient Health Questionnaire-9 (PHQ-9) over time | change from baseline (one week before the first session of PM+) to post assessment (one week after the last session of PM+); which is expected to last an average of 7 weeks
  PHQ-9 is a 9-item questionnaire that aims to measure the depressive symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day) providing a range between 0 and 27. Higher scores indicate more severe depressive symptoms.

SECONDARY OUTCOMES:
Change of the Generalized Anxiety Disorder-7 (GAD-7) over time | change from baseline (one week before the first session of PM+) to post assessment (one week after the last session of PM+); which is expected to last an average of 7 weeks
  GAD-7 is a 7-item measure of general anxiety symptoms that measures anxiety symptoms. Each item is scored from 0 (not at all) to 3 (nearly every day) providing a range between 0 and 21. Higher scores indicate higher levels of anxiety.
Change of the Posttraumatic Stress Disorder Checklist for Diagnostic and Statistical Manual-5 (DSM-5) (PCL-5) over time | change from baseline (one week before the first session of PM+) to post assessment (one week after the last session of PM+); which is expected to last an average of 7 weeks
  The PCL-5 is a 20-item questionnaire that assesses the symptoms of PTSD. Items are scored from 0 (not at all) to 4 (extremely) providing a range between 0 and 16. Higher scores indicate higher levels of PTSD symptoms.
Change of the Kessler Psychological Distress Scale (K-10) over time | change from baseline (one week before the first session of PM+) to post assessment (one week after the last session of PM+); which is expected to last an average of 7 weeks
  K-10 is a 10-item scale that assesses the psychological distress. Each item is scored from 1 (none of the time) to 5 (all of the time) and ranges between 10 and 50. Higher scores indicate more severe psychological distress.
Change of the World Health Organization Disability Assessment Schedule (WHODAS 2.0) over time | change from baseline (one week before the first session of PM+) to post assessment (one week after the last session of PM+); which is expected to last an average of 7 weeks
  WHODAS is a 12-item scale that assesses ability to engage in daily activities. Each item is scored from 0 (none) to 4 (extreme) and ranges between 0 and 48. Higher scores indicate more daily dysfunctioning.
Change of the the psychological outcomes profiles (PSYCHLOPS) over time | change from baseline (one week before the first session of PM+) to post assessment (one week after the last session of PM+); which is expected to last an average of 7 weeks
  PSYCHOLOPS is a scale that asks two problems and evaluates the level of distress about those problems on a 6-point scale (with higher scores indicating greater severity).

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Coşkun Toker, PhD student, Study Chair — Koç University
Locations (1):
- Koç University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Background] Sangraula M, Turner EL, Luitel NP, van 't Hof E, Shrestha P, Ghimire R, Bryant R, Marahatta K, van Ommeren M, Kohrt BA, Jordans MJD. Feasibility of Group Problem Management Plus (PM+) to improve mental health and functioning of adults in earthquake-affected communities in Nepal. Epidemiol Psychiatr Sci. 2020 May 26;29:e130. doi: 10.1017/S2045796020000414. PMID 32452336